CLINICAL TRIAL: NCT01562509
Title: Improvement of Hospital Care for Patients With Non-Hodgkin's Lymphoma
Brief Title: PEARL Study: Improvement of Non-Hodgkin's Lymphoma Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZonMW 171103002
Record Dates: First submitted 2012-03-08; First posted 2012-03-23 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Non-Hodgkin lymphoma (NHL); Quality of health care; Oncology Service Hospital; Patient-centredness; PROMs
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard implementation strategy (Active Comparator): Standard intervention
  Interventions: Other: Standard intervention
- Innovative implementation strategy (Experimental): Implementation tools
  Interventions: Other: Implementation tools

INTERVENTIONS:
Other: Implementation tools — * Professionals receive audit & feedback
  * Patients (and clinicians) have access to a website with information tailored to patients with an NHL. This website gives insight into the logistic processes of each diagnostic tool and into the patients' personal care pathway.
  * Standardization of diagnostic and evaluative request forms and reports for clinicians.
  * Supporting material for standardizing the procedure for multidisciplinary meetings.
  Arms: Innovative implementation strategy
Other: Standard intervention — Standard intervention consists of audit&feedback
  Arms: Standard implementation strategy

SUMMARY:
The main objective of the proposed study is to assess the effectiveness, feasibility and costs of a tailored strategy (developed in accordance with the barriers found and current practice) to improve care for patients with non-Hodgkin's lymphomas (NHL), compared to a common strategy of 'audit & feedback'.

DETAILED DESCRIPTION:
In a previous study among 22 Dutch hospitals many gaps in the care for patients with non-Hodgkin's lymphomas (NHL) were found, compared to best evidence as described in guidelines. In a problem analysis study, barriers and facilitators for good quality of NHL-care were assessed and a tailored implementation strategy was developed, based on these findings. The proposed study aims at the effectiveness, feasibility and costs of this tailored strategy to improve quality of care for patients with an NHL in a clustered randomized controlled trial in 19 Dutch hospitals.

Multilevel regression analyses will be performed to evaluate the effectiveness of both strategies. Exposure to and experiences with the strategy elements will be analysed descriptively.

Regarding the costs, the two strategies are compared with a health care perspective. The input of resources will be assessed by collecting volumes of consumed resources and multiplying these by the price of each resource unit; the implementation process and consequently costs will be estimated by an Activity Based Costing (ABC) approach. The output will be determined by the level of adherence to the NHL quality indicators.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-Hodgkin lymphoma
* Diagnosed in one of the participating hospitals
* Able to read and understand Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in adherence to quality indicators for NHL care | baseline and 1 year
  The effect of our interventions will be measured by means of adherence to quality indicators for optimal NHL care. The effects of the audit and feedback strategy (9 hospitals) versus the tailored strategy (9 hospitals) will be evaluated using previously developed quality indicators. These indicators for optimal NHL care were developed on the basis of evidence based guidelines, literature and opinions of clinicians about NHL care in a previous study and were validated.

SECONDARY OUTCOMES:
Exposure to and experiences with the interventions | after 1 year
  To study the feasibility of both strategies, a process evaluation has to give insight into the mechanisms and processes responsible for the result (= extent of adherence to the indicator set for optimal NHL care). The actual 'exposure' of the patients and professionals to the implementation elements, together with their experience with these elements may have influenced the final result (success or failure of adherence). Data about 'exposure' to the different interventions will be collected using questionnaires.
Costs of the strategy and the changed care | after 1 year
  Non-adherence to the multidisciplinary NHL guideline may lead to unnecessary medical interventions and more complications, and subsequently to efficiency losses. This economic evaluation compares the two implementation strategies. The perspective of this economic evaluation will be a health care perspective. Both the costs of the implementation strategy and changes in health care consumption will be assessed. The outcome should facilitate local health care decision making on implementation.
Change from baseline in morbidity | baseline and 1 year
  Morbidity is an important outcome measure for the effect of the intervention strategy.
Differences between both groups in Patient Related Outcome Measures (PROMs) | after 1 year
  Patient Related Outcome Measures as quality of life are important measures to evaluate the outcome of care from a patient perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Rosella Hermens, PhD, Principal Investigator — Radboud University Nijmegen Medical Center; Nelleke Ottevanger, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Stienen JJ, Hermens RP, Wennekes L, van de Schans SA, Dekker HM, Blijlevens NM, van der Maazen RW, Adang EM, van Krieken JH, Ottevanger PB. Improvement of hospital care for patients with non-Hodgkin's lymphoma: protocol for a cluster randomized controlled trial (PEARL study). Implement Sci. 2013 Jul 9;8:77. doi: 10.1186/1748-5908-8-77. PMID 23837833
- [Background] Stienen JJ, Ottevanger PB, Wennekes L, van de Schans SA, Dekker HM, Blijlevens NM, van der Maazen RW, van Krieken JH, Hermens RP. Delivering high-quality care to patients with a non-Hodgkin's lymphoma: barriers perceived by patients and physicians. Neth J Med. 2014 Jan;72(1):41-8. PMID 24457441